CLINICAL TRIAL: NCT06726759
Title: RELATIONSHIP BETWEEN FORWARD HEAD POSTURE and HAMSTRING TIGHTNESS in YOUNG ADULTS
Brief Title: RELATIONSHIP BETWEEN FORWARD HEAD POSTURE and HAMSTRING TIGHTNESS
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mark Refat Gabra Hana, mark refat gabra hana, Cairo University
Other Study IDs: FHP and hamstring tightness
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Forward Head Posture

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 50 males: 50 males with FHP and their BMI was between 20 and 25 kg/m2 ang ranged between 18 and 25 years
- 50 females: females with forward head posture and their BMI was between 20 and 25 kg/m2 and their age ranged between 18 and 25 years

SUMMARY:
The purpose of this study will be to investigate:

1. Relationship between forward head posture and hamstring tightness in young adults
2. The gender specific effect (female versus male) on the relationship between forward head posture and hamstring tightness in young adults

DETAILED DESCRIPTION:
Forward head posture imposes approximately 3.6 times more pressure on the neck than proper posture, and the prolonged burden of supporting the increased head weight can potentially cause neck pain, fatigue, and chronic musculoskeletal disorders. Hamstring tightness can cause posterior pelvic tilt, which leads to decreased lordosis of lumbar spine and resulting in LBP. Hamstring tightness can contribute to various issues, including muscle strains,loss of lumbar spine curvature, sacroiliac joint disorders, and plantar fasciitis. These problems primarily arise due to misalignment of the body and imbalanced force distribution between muscles and joints. Hamstring and sub-occipital muscles are connected by a neural system and sub-occipital muscles pass through the dura mater. this is called superficial back line (SBL), which connects the lower extremities, trunk, neck, and head protects the body's entire posterior surface and provides an important function of up-righting the body. There is still lack of research work about the relationship between FHP and hamstring muscle tightness and the gender-specific effect (female versus male) on the relationship between FHP and hamstring tightness in young adults.

ELIGIBILITY:
Inclusion Criteria:

* Both genders were included, with an age ranged between 18 and 25 years old.
* Participants with a CVA equal to or less than 49° were included (Haytham M. Elhafez, 2023).
* Body mass index was between 18 and 25 kg. /m2 (Haytham M. Elhafez, 2023).

Exclusion Criteria:

* Systemic disease
* History of hamstring injury within the last 2 years
* Previous knee injury
* Fracture in the spine or lower limb
* Spinal or lower limb surgery
* Pregnancy
* Congenital deformity
* Leg length discrepancy more than 2cm
* Acute spasm of hamstring muscles
* Neuromuscular disorders of the lower extremity, like stroke, muscular dystrophy and peripheral neuropathy
* History of any malignancy or infectious disease
* Spinal or limb deformities

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — males and females
Study Population: young adults with forward head posture
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
craniovertebral angle and hamstring flexibility angle | july -november 2024
  craniovertebral angle is the angle formed between a horizontal line through the spinous process of C7 and a line from the tragus of the ear craniovertebral angle was measured by Photogrammetry and kinovia software hamstring flexibility angle was measured by active knee extension test and kinovia software video analysis

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy, Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: this study compare the immediate effects of application of the suboccipital muscle inhibition and self-myofascial release techniques in the suboccipital region on short hamstring — https://pubmed.ncbi.nlm.nih.gov/25642072/